CLINICAL TRIAL: NCT03906851
Title: Effects of a School Based Health Promoting Intervention With Physical Activity and Nutrition Among 8th Graders in Telemark
Brief Title: Active and Healthy Kids in Telemark - a School Based Health Promoting Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South-Eastern Norway (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACTIKIDS
Record Dates: First submitted 2018-01-19; First posted 2019-04-08 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2022-10

CONDITIONS: Academic Performance; Physical Fitness; Physical Activity; Nutrition
Keywords: School; Health; Academic performance; Physical activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity and diet (Experimental): Multi-component, holistic model with a) physical activity, b) nutrition, and c) psychosocial work.
  A: physical activity will be provided as a pedagogical tool in subjects Mathematics, Norwegian and English B: Focus on school meals and menus in school cafeteria C: Psychosocial work with focus on the associations between physical activity, nutrition and psychosocial health. Collaboration between schools and school health services
  Interventions: Behavioral: Activity and diet
- Control (No Intervention): Schools are required to perform teaching activities, school meals and school cafeteria menus as usual

INTERVENTIONS:
Behavioral: Activity and diet — Physical activity: use of physical activity in theoretical subjects (3 x 30 min/week), physically active breaks (5 x 5 min/week), physical education (2 x 45 min/week) Nutrition: focus on school meals
  Arms: Activity and diet

SUMMARY:
The study examine possible changes in physical activity, nutrition, and psychosocial health following the intervention "Active and Healthy Kids in Telemark". The intervention schools will received the intervention, whereas the control schools will continue as usual.

DETAILED DESCRIPTION:
School based, health promoting interventions with focus on increase physical activity and improved nutrition seems to be a good solution to the challenges with low physical activity level, poor physical fitness, poor nutrition and psychosocial health challenges among children and adolescents. Low physical activity levels and physical fitness is recognized as one of the major public health challenges in the 21st century, and it negatively affects cognitive skills and academic performances. Providing school based health promoting interventions makes it easier to reach all children and adolescents regardless of social and cultural background, and hence reduce social inequalities in health.

ELIGIBILITY:
Inclusion Criteria:

* Pupil 8th grade

Exclusion Criteria:

* Inadequate language skills to complete questionnaire

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 840 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Physical activity (counts per minute) | 4 days
  Objectively assessment of physical activity by accelerometer Actigraph GT3x

SECONDARY OUTCOMES:
Physical fitness: Andersen test | 10 minutes
  Andersen test to measure endurance capacity, running test on 20 m track for 10 minutes. Number of metres ran during the 10 minutes is registered.
Physical fitness: standing long jump | 2 minutes
  Standing long jump to measure explosive strength. Each subject gets two trials. Longest trial is registered in cm.
Nutrition and diet: questionnaire | 5 minutes
  self-report through own-developed questionnaire (not standardised scale)
Health-related Quality of Life | 10 minutes
  KIDSCREEN-27 (unabbreviated name) is a 27 item self-report instrument for health-related quality of life in children and adolescents. Each item is scored on a Likert scale from 1 to 5. The scores of each item are clustered into five dimensions: Physical Well-Being, Psychological Well-Being, Autonomy & Parents, Peers & Social Support and School Environment. Each dimension, or subscale, is scored as Rasch scales (i.e., sum of item scores for each subscale, transform the raw sumscores into Rasch person parameter estimates and T-values according to the KIDSCREEN-27 manual (KIDSCREEN group Europe, 2006)). For all these dimensions, higher Rasch scores and T-scores indicate better quality of life according to that given dimension.
Academic performance: grades in subjects Norwegian, mathematics and English | 45 minutes
  Results from national tests which assess level of academic performance among the pupils

CONTACTS AND LOCATIONS:
Overall Officials: Solfrid Bratland-Sanda, PhD, Study Chair — University College of Southeast Norway
Locations (1):
- University College of Southeast Norway, Bø, Telemark, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naylor PJ, Nettlefold L, Race D, Hoy C, Ashe MC, Wharf Higgins J, McKay HA. Implementation of school based physical activity interventions: a systematic review. Prev Med. 2015 Mar;72:95-115. doi: 10.1016/j.ypmed.2014.12.034. Epub 2015 Jan 6. PMID 25575800
- [Background] Mura G, Vellante M, Nardi AE, Machado S, Carta MG. Effects of School-Based Physical Activity Interventions on Cognition and Academic Achievement: A Systematic Review. CNS Neurol Disord Drug Targets. 2015;14(9):1194-208. doi: 10.2174/1871527315666151111121536. PMID 26556088
- [Background] Ho FK, Louie LH, Chow CB, Wong WH, Ip P. Physical activity improves mental health through resilience in Hong Kong Chinese adolescents. BMC Pediatr. 2015 Apr 22;15:48. doi: 10.1186/s12887-015-0365-0. PMID 25898349
- [Background] Penedo FJ, Dahn JR. Exercise and well-being: a review of mental and physical health benefits associated with physical activity. Curr Opin Psychiatry. 2005 Mar;18(2):189-93. doi: 10.1097/00001504-200503000-00013. PMID 16639173
- [Background] Ravens-Sieberer, U. and K.G. Europe, The Kidscreen Questionnaires: Quality of Life Questionnaires for Children and Adolescents ; Handbook. 2006: Pabst Science Publ.
- [Derived] Bratland-Sanda S, Schmidt SK, Reinboth MS, Vrabel KA. Under pressure to exercise: a cross-sectional study of characteristics and predictors of compulsive exercise in early adolescents. J Eat Disord. 2022 Nov 5;10(1):156. doi: 10.1186/s40337-022-00686-8. PMID 36335366